# Janssen Research & Development Biostatistics and Programming

# Statistical Analysis Plan/Data Presentation Specifications for Clinical Study Report

A Randomized, Open-label, Multicenter, Multiphase Study of JNJ-63723283, an Anti-PD-1 Monoclonal Antibody, Administered in Combination with Daratumumab, Compared with Daratumumab Alone in Subjects with Relapsed or Refractory Multiple Myeloma

Protocol 54767414MMY2036; Phase 2/3 JNJ-63723283; JNJ-54767414 (DARZALEX®, daratumumab)

Date: 25 September 2018

**Status:** Approved

Date: 25 September 2018

**Prepared by:** Janssen Research & Development, LLC

**Document No.:** EDMS-ERI-167849379:2.0

**Compliance:** The study described in this report was performed according to the principles of Good Clinical Practice (GCP).

### **Confidentiality Statement**

The information in this document contains trade secrets and commercial information that are privileged or confidential and may not be disclosed unless such disclosure is required by applicable law or regulations. In any event, persons to whom the information is disclosed must be informed that the information is privileged or confidential and may not be further disclosed by them. These restrictions on disclosure will apply equally to all future information supplied to you that is indicated as privileged or confidential.

# **TABLE OF CONTENTS**

| TAB | BLE OF CONTENTS | 2 |
|------------|-----------------------------------------------------------|----|
| LIST | T OF IN-TEXT TABLES AND FIGURES | 2 |
| AME | ENDMENT HISTORY | 3 |
| 1. | ANALYSIS DETAILS | |
| 1.<br>1.1. | | |
| 1.1. | | |
| 1.3. | | |
| 1.4. | | |
| 1.5. | | |
| 1.6. | Efficacy | 7 |
| 1.7. | | |
| 1.8. | | 8 |
| 1.9. | Biomarker | 9 |
| <b>2</b> . | LIST OF PLANNED OUTPUT | 10 |
| 3. | COLUMN LAYOUTS FOR TABLES | 15 |
| 4. | MOCK LAYOUTS | |
| <b>5</b> . | NARRATIVE CRITERION | 49 |
| 6. | PROGRAMMING CODE FOR STATISTICAL PROCEDURES (IF REQUIRED) | 49 |
| <b>7</b> . | LIST OF POST HOC OUTPUT (IF REQUIRED) | 49 |
| 8. | ADDITIONAL ANALYSIS/DEVIATION RULES | 49 |
| REF | FERENCES | 50 |
| LIS | T OF IN-TEXT TABLES AND FIGURES | |
| TAI | BLES | |
| Tabl | le 1: Demographic Variables | 6 |
| | le 2: Baseline Disease Characteristics | |
| FIG | GURES | |
| Fiau | ure 1: Study Scheme | 4 |

# **AMENDMENT HISTORY**

The statistical analysis plan (SAP) has been revised and description of the changes and the section affected are provided below.

| <b>Amendment -1</b> (07Sep2018) |
|---------------------------------------------------|
| Summary of change: 1. Included biomarker analysis |

| Applicable Section | Description of Change |
|---|---|
| 1.9 Biomarker | Since biomarker analysis would be included in the final CSR, this new section for biomarker analysis was added in this SAP. |

### 1. ANALYSIS DETAILS

This document contains definitions of analysis sets, derived variables and planned data presentation specifications which will be used in clinical study report of study 54767414MMY2036. The analysis will be performed after final data base lock when protocol 54767414MMY2036, Amendment 2 is approved and implemented at all sites.

# 1.1. Overview of Study Design

This is a randomized, open-label, multicenter, multiphase study assessing the efficacy and safety of JNJ-63723283 (an anti-PD-1 monoclonal antibody) in combination with daratumumab compared with daratumumab alone in subjects with multiple myeloma who have received at least 3 prior lines of therapy including a PI and an IMiD or whose disease is double refractory to both a PI and an IMiD. A diagram of the study design is provided in Figure 1.





As of 25 May 2018, the Sponsor terminated further enrollment into this study and subjects in Screening were deemed Screen Failures and were not further randomized into the study. Subjects continuing on study will receive daratumumab monotherapy starting 25 May 2018. Part 3 is no longer applicable for this study.

# 1.2. Analysis Sets

- Safety analysis set: includes all subjects who have received at least 1 dose of study agent (JNJ-63723283 or daratumumab, partial or complete) in either Safety Run-in Part 1 or Part 2 of the study. This analysis set will be used for below analyses.
- Pharmacokinetics (PK)-evaluable analysis set: includes all subjects who have received at least 1 dose of daratumumab or JNJ-63723283 and have at least 1 post-infusion sample in Safety Run-in Part 1 of the study.
- Immunogenicity analysis set: include all subjects who have received at least 1 dose of JNJ-63723283 or daratumumab and have appropriate serum samples for detection of antibodies to JNJ-63723283 or daratumumab (i.e., subjects with at least 1 sample obtained after their first dose of JNJ-63723283 or daratumumab) in Safety Run-in Part 1 of the study.

# 1.3. Treatment Groups

The treatment groups are Safety Run-in (JNJ-63723283+daratumumab); and Arm A (daratumumab alone) and Arm B (JNJ-63723283+ daratumumab) for Part 2.

## 1.4. End of Follow-up and Duration of Follow-up

The end of follow-up is the date of death for subjects who died. For those who are still alive, the end of follow-up is defined as the maximum date of the following study evaluations: labs (hematology, chemistry, serology, coagulation, thyroid function), adverse events, vital signs, ECOG performance status, study drug administration, 12-lead ECG, pre-infusion medications, post-infusion medications, concomitant medications, subsequent anti-cancer treatment, tumor assessment, clinical events/disease response per investigator and date of last known to be alive.

Duration of follow-up (in months) equals the end of follow-up minus the first dosing date plus 1 for Part 1 and equals the end of follow-up minus the randomization date plus 1 for Part 2, divided by 365.25/12.

Study duration of follow-up will be summarized by treatment group and overall for safety Analysis Set.

# 1.5. Subject information

The distribution of subjects by region and country will be presented for safety analysis set by treatment group and overall.

• **Demographics and baseline characteristics:** Demographics and baseline characteristics will be summarized for safety analysis set by treatment group and overall. A listing of subject demographic and baseline characteristics will be provided as well. Table 1 and Table 2

respectively present a list of the demographic variables and baseline disease characteristics that will be summarized by treatment group and overall.

**Table 1: Demographic Variables** 

| Continuous Variables: | Summary Type |
|---|---|
| Age (years) | Descriptive statistics (N, mean, |
| Weight (kg) | standard deviation [STD], median |
| Height (cm) | and range [minimum and |
| | maximum]). |
| Categorical Variables | |
| Age ( $<65$ years, $\ge65$ years and $<75$ years, $\ge75$ years) | |
| Weight (≤65kg, >65kg and ≤85kg, >85kg) | |
| Sex (male, female) | N, frequency distribution with the |
| Race (American Indian or Alaska Native, Asian, Black or African | number and percentage of |
| American, Native Hawaiian or other Pacific Islander, White, | subjects in each category. |
| Multiple <sup>a</sup> , not reported) | subjects in each category. |
| Ethnicity (Hispanic or Latino, not Hispanic or Latino, not reported) | |
| Baseline ECOG (0, 1, 2) | |

<sup>&</sup>lt;sup>a</sup> If multiple race categories are indicated, the Race is recorded as 'Multiple'

**Table 2: Baseline Disease Characteristics** 

| Continuous Variables: | Summary Type |
|---|---|
| Time since MM diagnosis (years) | Descriptive statistics (N, mean, |
| | standard deviation [STD], median |
| | and range [minimum and |
| | maximum]). |
| Categorical Variables | |
| Type of multiple myeloma (IgG, IgA, IgM, IgD, IgE, light | |
| chain only [kappa and lambda], biclonal, negative | |
| immunofixation, not detected) | |
| Type of measurable disease (serum measurable only [IgG, IgA | |
| and Other], both serum and urine measurable, urine measurable | |
| only, serum FLC measurable) | |
| ISS staging at screening by central laboratory assessment (I, II, | |
| III) | N, frequency distribution with the |
| Number of lytic bone lesions (None, 1-3, 4-10, more than | number and percentage of subjects |
| 10) | in each category. |
| Presence of diffuse myeloma-related osteopenia (Yes, No) | |
| Number of extramedullary plasmacytomas $(0, \ge 1)$ | |
| Bone marrow % plasma cells (<10, 10 – 30, >30) | |
| Status of cytogenetic abnormality (standard-risk, high-risk | |
| [Del17p, T(4;14), T(14;16)]), | |
| ECG overall conclusion (normal, abnormal [clinically | |
| significant, not clinically significant, not evaluable) | |

• **Subject Disposition:** The number of subjects in the following disposition categories will be summarized throughout the study for safety population by treatment group and overall: subjects who discontinued study treatment, reasons for discontinuation of study treatment, subjects who terminated study prematurely, and reasons for termination of study. Listings of subjects will be provided for the following categories: subjects who discontinued study treatment, and subjects who terminated study prematurely.

- **Medical history:** Medical history collected at baseline or screening visit will be summarized by system-organ class and preferred term for each treatment group and overall.
- **Prior and concomitant medication:** Summaries of concomitant medications will be presented by therapeutic class, pharmacologic class and preferred term by treatment group and overall for safety population. A summary of prior therapies (systemic therapy, radiotherapy, or cancer-related surgery/ procedure) will be provided by treatment group. Specifically, the number of prior lines of therapy will be calculated according to IWMG consensus guidelines (Durie 2006; Kumar 2016; Rajkumar 2011) <sup>1,2,3</sup> and summarized by the following categories: ≤ 3 and > 3 through frequency and descriptive statistics. Subjects with prior cancer-related surgery/procedure and with prior radiotherapy will be listed for safety population.
- **Pre-infusion and post-infusion medication:** Pre-infusion and post-infusion medication will be summarized by therapeutic class, pharmacologic class and preferred term by treatment group and overall for safety population. A listing will be provided for pre-infusion medication and post-infusion medication, respectively.
- Exposure: Summary of treatment exposure will be provided for safety population. The total number of treatment cycles received for each subject will be summarized by frequency and descriptive statistics (N, mean [SD], median, range [minimum, maximum]) by treatment group. Descriptive statistics for duration of study treatment, defined as (date of last dose of study treatment date of first dose of study treatment) +1, will be presented by treatment group. Subject-month of exposure are calculated as days of duration/365.25\*12. Total number of daratumumab and JNJ-63723283 infusions will be calculated. respectively. Exposure will be listed for safety population.

The number and percentage of subjects with treatment cycle delay will be calculated by treatment group. The frequencies of actions planned prior to infusion start (infusion delayed, infusion skipped or study drug permanently discontinued) and taken during infusion (infusion interrupted, infusion rate decrease, infusion aborted) will be summarized, together with reasons reported (adverse events or other) accordingly.

Descriptive statistics will be presented for the following parameters: dose and relative dose intensity of daratumumab, dose and relative dose intensity of JNJ-63723283.

• **Protocol deviation:** A listing of subjects with major protocol deviations including treatment group, subject ID, type of deviation, and reasons for deviation will be provided.

# 1.6. Efficacy

A listing of subjects' best response, and disease progressions based on investigator's assessment, and overall survival will be provided for the safety analysis set, including treatment group, subject ID, and baseline measurable disease type. For subjects who had progression disease (PD), the PD reasons based on investigator's assessment will be listed.

# 1.7. Safety

#### • Adverse events:

- An overview of treatment-emergent adverse events (TEAEs) will be summarized for safety population by treatment group and overall.
- Incidence of TEAEs will be summarized by MedDRA SOC, and preferred term.
- List of subjects with any TEAEs, serious TEAEs, toxicity grade 3 or 4 TEAEs, treatmentemergent Infusion Related Reactions (IRRs), and immune-mediated TEAEs will be provided for safety population.
- List of subjects with any TEAEs leading to all treatment discontinuation, TEAEs leading to any treatment discontinuation, TEAEs with outcome death, TEAEs leading to cycle delay or dose modifications, and TEAEs leading to infusion interrupted, infusion rate decreased or infusion aborted will be provided for safety population.
- Subjects who died during the study, and had new malignancies will also be listed, respectively.
- Laboratory values: Laboratory values will be listed at each time points for safety analysis set.
  - The hematology parameters include: hemoglobin, lymphocytes, neutrophils, platelet, and white blood cell (WBC).
  - The chemistry parameters include: alanine aminotransferase (ALT), alkaline phosphatase, aspartate aminotransferase (AST), amylase, calcium, creatinine, creatinine clearance, potassium, sodium, total bilirubin, and total lipase,
  - The thyroid function parameters include: free thyroxine, free triiodothyronine, thyroid stimulating hormone, and total triiodothyronine.
- **Electrocardiograms (ECG):** ECG values will be reported at each time points for safety analysis set in listings.
- **Vital signs:** Vital signs will be listed at each time points for safety analysis set. The variables include: weight, blood pressure (systolic and diastolic).

# 1.8. Pharmacokinetics/Immunogenicity

- **Pharmacokinetics:** PK analyses will be performed on the PK-evaluable population. The pharmacokinetic parameters are defined as
  - Minimum observed concentration (C<sub>min</sub>) the concentration observed immediately before infusion.
  - Maximum observed concentration (C<sub>max</sub>) the concentration observed after the end of infusion

For both JNJ-63723283 and daratumumab, the PK evaluations include  $C_{min}$  and  $C_{max}$ . All serum concentrations below the lowest quantifiable concentration or missing data will be labeled as such in the concentration data presentation. Concentrations below the lowest quantifiable concentration will be treated as zero in the summary statistics.

The  $C_{min}$  and  $C_{max}$  will be summarized at each sampling time point by descriptive statistics (N, mean, STD, median, range, coefficient variation and geometric mean) for JNJ-63723283 and daratumumab, respectively, by treatment group. Line plot of mean ( $\pm$ STD) daratumumab and JNJ-63723283 serum peak and trough concentrations over time will be provided.

• Immunogenicity: Immunogenicity analyses will be performed on the immunogenicity analysis set. The incidence of anti-daratumumab and anti-JNJ-63723283 antibodies will be summarized for all subjects who receive a dose of daratumumab or JNJ-63723283 and have appropriate samples for detection of antibodies to daratumumab or JNJ-63723283 by treatment group. In addition, subjects who are positive for antibodies to daratumumab or JNJ-63723283 will also be listed.

## 1.9. Biomarker

Descriptive statistics for values and changes from baseline at each scheduled visit for absolute counts (cells/µl) and percentage of total NK cells, CD8+ T cells, and B cells in peripheral blood will be provided by treatment group. Similar analysis for total and CD38+ myeloid derived suppressor cells (MDSCs), and total and CD38+ regulatory T cells (Tregs) will be performed. Plots for these biomarkers over time will be provided. In additional, percent of activated CD8+ T cells will be summarized and plotted.

# 2. LIST OF PLANNED OUTPUT

| Output<br>Identifier | Output Title | Analysis Set | Use for<br>What Effort<br>(TLR, IA,<br>INTXT,<br>DMC) | Reference<br>Mock | Column<br>Layout |
|---|---|---|---|---|---|
| Subject and Tr | eatment Information (SI) | | Direcy | 1 | |
| Subjec | t Disposition and Study Comple | tion/Withdrawal Int | formation | | |
| TSIDS01 | Subjects Disposition | Safety | INTXT | TSIDS-ST02 | 1 |
| LSIDS01 | Listing of Subjects Disposition | Safety | | LSIDS-ST01 | |
| TSIFU01 | Summary of Study Duration of Follow-up | Safety | INTXT | TSIFU01 | 1 |
| | raphics and Baseline Character | | | | |
| TSIPOP01 | Subject Populations for Evaluation | Safety | INTXT | TSIDEM-ST03 | 1 |
| TSIENR01 | Subject Enrollment by Region and Country | Safety | | TSIDEM-ST04 | 1 |
| TSIDEM01 | Summary of Demographics and Baseline Characteristics | Safety | INTXT | TSIDEM-ST01 | 1 |
| TSIDEM02 | Summary of Baseline Disease Characteristics; | Safety | INTXT | TSIDEM02 | 1 |
| LSIDEM01 | Listing of Demographics and Baseline Characteristics | Safety | | LSIDEM-ST01 | |
| TSIMH01 | Summary of Medical History<br>by MedDRA System Organ<br>Class and Preferred Term | Safety | | TSIMH01 | 1 |
| | and Concomitant Therapies | | | | |
| TSIPM01 | Summary of Prior Systemic<br>Therapy | Safety | INTXT | TSIPM01 | 1 |
| TSICM01 | Summary of Concomitant<br>Medications | Safety | | TSICM-ST01 | 1 |
| TSICM02 | Summary of Pre-infusion<br>Medications | Safety | | TSICM-ST01 | 1 |
| TSICM03 | Summary of Post-infusion<br>Medications | Safety | | TSICM-ST01 | 1 |
| LSICM01 | Listing of Pre-infusion Medications | Safety | | LSICM01 | |
| LSICM02 | Listing of Post-infusion<br>Medications | Safety | | LSICM02 | |
| LSIPM01 | Listing of Subjects with Prior<br>Cancer-related<br>Surgery/Procedure | Safety | | LSIPM01 | |
| LSIPM02 | Listing of Subjects with Prior<br>Radiotherapy | Safety | | LSIPM02 | |
| | ol Deviations | | | | |
| LSIDEV01 | Listing of Subjects with Major<br>Protocol Deviations | Safety | | LSIDEV-ST01 | |
| | of Exposure | Laga | T | Lagrant: | 1 - |
| TSIEXP01 | Summary of Treatment<br>Cycles, Duration of Study<br>Treatment and Dose Intensity | Safety | INTXT | TSIEX-ST01 | 2 |

Statistical Analysis Plan/Data Presentation Specifications 54767414MMY2036

| Output<br>Identifier | Output Title | Analysis Set | Use for<br>What Effort<br>(TLR, IA,<br>INTXT,<br>DMC) | Reference<br>Mock | Column<br>Layout |
|---|---|---|---|---|---|
| TSIEXP02 | Summary of Treatment Cycle<br>Delays, Incidences of and<br>Reasons for Study Treatment<br>Dose Modifications | Safety | | TSIEXP02 | 2 |
| TSIEXP03 | Summary of Action Taken During the Infusion | Safety | | TSIEXP03 | 2 |
| LSIEX01 | Listing of Treatment Exposure | Safety | | LSIEX-ST01 | |
| Efficacy Result | (FF) | | | | |
| LEFRSP01 | Listing of Efficacy Variables Based on Investigator Assessment | Safety | | LEFRSP01 | |
| Safety Results | (CF) | | | | |
| | se Events | | | | |
| TSFAE01 | Overview of Treatment-<br>emergent Adverse Events | Safety | INTXT | TSFAE-ST01 | 1 |
| TSFAE02 | Treatment-emergent Adverse<br>Events by System Organ<br>Class and Preferred Term | Safety | INTXT | TSFAE-ST02 | 1 |
| LSFAE01 | Listing of Treatment-emergent<br>Adverse Events | Safety | | LSFAE01 | |
| LSFAE02 | Listing of Treatment-emergent<br>Serious Adverse Events | Safety | | LSFAE01 | |
| LSFAE03 | Listing of Treatment-emergent<br>Grade 3 or 4 Adverse Events | Safety | | LSFAE01 | |
| LSFAE04 | Listing of Subjects who Discontinued All Study Treatment Because of 1 or More Treatment-emergent Adverse Events; | Safety | | LSFAE01 | |
| LSFAE05 | Listing of Subjects Who Discontinued Any of Study Drugs Because of 1 or More Treatment-emergent Adverse Events | Safety | | LSFAE01 | |
| LSFAE06 | Listing of Treatment-emergent<br>Infusion Related Reactions | Safety | | LSFAE01 | |
| LSFAE07 | Listing of Immune-mediated<br>Treatment-emergent Adverse<br>Event | Safety | | LSFAE01 | |
| LSFAE08 | Listing of Treatment-emergent<br>Adverse Events Leading to<br>Cycle Delay or Dose<br>Modifications | Safety | | LSFAE01 | |
| LSFAE09 | Listing of Treatment-emergent<br>Adverse Events Leading to<br>Infusion Interrupted, Infusion<br>Rate Decreased or Infusion<br>Aborted | Safety | | LSFAE01 | |

| Output<br>Identifier | Output Title | Analysis Set | Use for<br>What Effort<br>(TLR, IA,<br>INTXT,<br>DMC) | Reference<br>Mock | Column<br>Layout |
|---|---|---|---|---|---|
| LSFAE10 | Listing of Subjects Who Had<br>New Malignancies | Safety | | LSFAE10 | |
| LSFDTH01 | Listing of Subjects Who Died<br>During the Study | Safety | | LSFDTH-ST01 | |
| Clinical L | <br>aboratory Evaluation | | | | |
| TSFLAB01 | Shift Table of Baseline versus Worst Toxicity Grade during Treatment in Hematological Test | Safety | | TSFLAB-ST07 | 2 |
| TSFLAB02 | Shift Table of Baseline versus<br>Worst Toxicity Grade during<br>Treatment in Biochemistry<br>Test; | Safety | | TSFLAB-ST07 | 2 |
| LSFLAB01 | Listing of Other Laboratory<br>Values | Safety | | LSFLAB-ST01 | |
| Electrocard | iograms | | | | |
| LSFECG01 | Listing of ECG Results | Safety | | LSFECG-ST01 | |
| Vital Signs | Eisting of Led Results | Buiety | | LSI LCG 5101 | ı |
| LSFVS01 | Listing of Vital Signs Values | Safety | | LSFLAB-ST01 | |
| Pharmacokinet | ics/Immunogenicity (PK/IR) | | | | |
| TPKCONC01 | Summary of Daratumumab Concentration (ug/mL) | PK-evaluable | INTXT | TPK-ST07 | 3 |
| TPKCONC02 | Summary of JNJ-63723283<br>Concentration (ug/mL) | PK-evaluable | INTXT | TPK-ST07 | 3 |
| GPKCONC01 | Mean (SD) Daratumumab<br>Serum Peak and Trough<br>Concentrations (ug/mL) | PK-evaluable | | GPK-ST05 | |
| GPKCONC02 | Mean (SD) JNJ-63723283<br>Serum Peak and Trough<br>Concentrations (ug/mL) | PK-evaluable | | GPK-ST05 | |
| TPKIR01 | Summary of Anti-<br>daratumumab Antibodies<br>Status | Immunogenicity | INTXT | TPKIR-ST01 | 4 |
| TPKIR02 | Summary of Anti-JNJ-<br>63723283 Antibodies Status | Immunogenicity | INTXT | TPKIR-ST01 | 4 |
| LPKCONC01 | List of Subjects Positive for<br>Anti-daratumumab Antibodies<br>Status | Immunogenicity | | LPKIR-ST01 | |
| LPKCONC02 | List of Subjects Positive for<br>Anti-JNJ-63723283<br>Antibodies Status | Immunogenicity | | LPKIR-ST01 | |
| Biomarkers | OH AHA CH | | | | |
| Natural K<br>TBMKNK01 | Summary of Percent of Total Natural Killer Cells in Blood | Safety | | TBMK01 | |
| | Over Time | | | | |

| Output<br>Identifier | Output Title | Analysis Set | Use for<br>What Effort<br>(TLR, IA,<br>INTXT,<br>DMC) | Reference<br>Mock | Column<br>Layout |
|---|---|---|---|---|---|
| TBMKNK02 | Summary of Total Natural<br>Killer Cells (Absolute Count)<br>in Blood Over Time | Safety | | TBMK01 | |
| GBMKNK01 | Plot of Percent of Total<br>Natural Killer cells in Blood<br>over time | Safety | | GBMK01 | |
| GBMKNK02 | Plot of Total Natural Killer<br>Cells (Absolute Count) in<br>Blood Over Time | Safety | | GBMK01 | |
| T Cells | | | | | |
| TBMKTC01 | Summary of Percent of CD8+<br>T Cells in Blood Over Time | Safety | | TBMK01 | |
| TBMKTC02 | Summary of CD8+ T Cells<br>(Absolute Count) in Blood<br>Over Time | Safety | | TBMK01 | |
| GBMKTC01 | Plot of Percent of CD8+ T<br>Cells in Blood Over Time | Safety | | GBMK01 | |
| GBMKTC02 | Plot of CD8+ T Cells<br>(Absolute Count) in Blood<br>Over Time | Safety | | GBMK01 | |
| TBMKTC03 | Summary of Percent of<br>Activated CD8+T Cells in<br>Blood Over Time | Safety | | TBMK01 | |
| GBMKTC03 | Plot of Percent of Activated<br>CD8+ T cells in Blood Over<br>Time | Safety | | GBMK01 | |
| B Cells | | • | | | |
| TBMKBC01 | Summary of Percent of B<br>Cells in Blood Over Time | Safety | | TBMK01 | |
| TBMKBC02 | Summary of B Cells<br>(Absolute Count) in Blood<br>Over Time | Safety | | TBMK01 | |
| GBMKBC02 | Plot of B Cells (Absolute<br>Count) in Blood Over Time | Safety | | GBMK01 | |
| GBMKBC01 | Plot of Percent of B Cells in<br>Blood Over Time | Safety | | GBMK01 | |
| CD38+ M | | | | | |
| TBMKMDSC<br>01 | Summary of Percent of Total<br>monocytic MDSCs in Blood<br>Over Time | Safety | | TBMK01 | |
| TBMKMDSC<br>02 | Summary of Percent of<br>CD38+ monocytic MDSCs in<br>Blood Over Time | Safety | | TBMK01 | |
| GBMKMDSC<br>01 | Plot of Percent of Total<br>monocytic MDSCs in Blood<br>over time | Safety | | GBMK01 | |
| GBMKMDSC<br>02 | Plot of Percent of CD38+<br>monocytic MDSCs in Blood<br>Over Time | Safety | | GBMK01 | |

Statistical Analysis Plan/Data Presentation Specifications 54767414MMY2036

| Output<br>Identifier | Output Title | Analysis Set | Use for<br>What Effort<br>(TLR, IA,<br>INTXT,<br>DMC) | Reference<br>Mock | Column<br>Layout |
|---|---|---|---|---|---|
| TBMKMDSC<br>03 | Summary of Total Monocytic<br>MDSCs (Absolute Count) in<br>Blood Over Time | Safety | | TBMK01 | |
| GBMKMDSC<br>03 | Plot of Total monocytic<br>MDSCs (Absolute Count) in<br>Blood Over Time | Safety | | GBMK01 | |
| CD38+ Tr | egs | • | • | • | · |
| TBMKTR01 | Summary of Percent of Total<br>Tregs in Blood Over Time | Safety | | TBMK01 | |
| TBMKTR02 | Summary of Percent of<br>CD38+ Tregs in Blood Over<br>Time | Safety | | TBMK01 | |
| TBMKTR03 | Summary of Total Tregs<br>(Absolute Count) in Blood<br>Over Time | Safety | | TBMK01 | |
| TBMKTR04 | Summary of CD38+ Tregs<br>(Absolute Count) in Blood<br>Over Time | Safety | | TBMK01 | |
| GBMKTR01 | Plot of Percent of Total Tregs in Blood Over Time | Safety | | GBMK01 | |
| GBMKTR02 | Plot of Percent CD38+ Tregs<br>in Blood Over Time | Safety | | GBMK01 | |
| GBMKTR03 | Plot of Total Tregs (Absolute Count) in Blood Over time | Safety | | GBMK01 | |
| GBMKTR04 | Plot of CD38+ Tregs<br>(Absolute Count) in Blood<br>Over Time | Safety | | GBMK01 | |

14

## 3. COLUMN LAYOUTS FOR TABLES

All tables listed in Section 2 are to be presented with the following columns layout, unless specified otherwise.

Layout 1: To be used in demographics, baseline disease characteristics, prior systemic therapies, medical history, TEAE overview, safety.

| Safety Run-in | Phase 2 | Total |
|---------------|---------|-------|
| | Arm A | |

Layout 2: To be used in exposure tables.

| Safety Run-in | Phase 2 |
|---------------|---------|
| | Arm A |

Layout 3: To be used in PK tables

| Safety Run-in | |
|---------------|-----------|
| Pre-dose | Post-dose |

Layout 4: To be used in immunogenicity tables



## Programming notes:

1. Footnotes that correspond to the naming of the treatment groups are specified as below: Key: Arm A = daratumumab alone;

## 4. MOCK LAYOUTS

TSIDS-ST02: Subjects Disposition; Safety Analysis Set (Study 54767414MMY2036)

| Analysis set: Safety | ### | ### | ### | ### | ### |
|---|---|---|---|---|---|
| Subjects who discontinued treatment<br>Reason for discontinuation | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Adverse Event | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Death | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Non-compliance with study drug | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Physician decision | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Pregnancy | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Progressive disease | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Study terminated by sponsor | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Subject refused further study | , | , , | , , | ` , | , |
| treatment | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Other | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ## (xx.x%) |
| Subjects who discontinued study<br>Reason for discontinuation | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Death | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Lost to follow-up | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Physician desicion | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Pregnancy | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Screen failure | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Study terminated by sponsor | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Withdrawal by subject | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Other | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |

Note: Percentages calculated with the number of subjects in each group as denominator.

| Display Specifications | |
|------------------------|---------|
| Output Identifier | TSIDS01 |

Programming Notes:

- 1. Reasons for discontinuation should be presented in descending frequency in the overall total column.
- 2. Remove the specific reason for discontinuation if there is no subject belongs to that.

## LSIDS-ST01: Listing of Subjects Disposition; Safety Analysis Set (Study 54767414MMY2036)

| | | | | Study Day <sup>a</sup> of Last | Total Dose for | Discontinuation | <u>1</u> |
|---|---|---|---|---|---|---|---|
| | | Subject | Disposition | Study Agent | Dara/JNJ283 | <u>Date</u> | Primary Reason for |
| Treatment Group | Site ID | ID | Event | Administered | (mg/kg or mg)b | (Study Day <sup>a</sup> ) | Discontinuation |

## **Display Specifications**

Output Identifier LSIDS01

Programming Notes:

- 1. Sort listing based on treatment group (Safety run-in, Arm A, Arm B), site ID, and subject ID.
- 2. Study day of last study agent administered is the study day that the subject received their last non-zero dose of study agent.
- 3. If the reason for discontinuation is Adverse event or Other, specify the AE preferred term or other reason in parentheses.

### TSIFU01: Summary of Study Duration of Follow-up; Safety Analysis Set (Study 54767414MMY2036)

| Analysis set: Safety | ## | ## | ## |
|--------------------------------|--------------|--------------|--------------|
| Duration of follow-up (months) | | | |
| N | ## | ## | ## |
| Mean (SD) | ##.# (##.##) | ##.# (##.##) | ##.# (##.##) |
| Median <sup>a</sup> | ## | ## | ## |
| Range | (##; ##) | (##; ##) | (##; ##) |

<sup>&</sup>lt;sup>a</sup> Based on Kaplan-Meier product limit estimate.

Note: Duration of follow-up is relative to the date of first dose.

### Programming Notes:

1. Mark '+" for the range values if come from the subjects who died, and the following footnote is needed: "+ Denotes subjects who died".

<sup>&</sup>lt;sup>a</sup> Study day is relative to the date of first dose of study agent.

<sup>&</sup>lt;sup>b</sup> Total dose is defined as a cumulative sum of all study agent administered. <u>Dara=daratumumab</u>; JNJ283=JNJ-63723283.

| TSIDEM-ST04: | Subject Enrollment by Region and Country; Safety Analysis Set (Study |
|---|---|
| | 54767414MMY2036) |

| Analysis set: Safety | ### | ### | ### | ### | ### |
|---|---|---|---|---|---|
| Region/Country | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Region 1 | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Country 1 | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Country 2 | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Country 3 | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |

Note: Percentages are calculated with the number of subjects in each group as denominator.

### Programming Notes:

1. Region and Country are presented in alphabetical order

TSIDEM-ST03: Subject Populations for Evaluation; Safety Analysis Set (Study 54767414MMY2036)

| Safety analysis set <sup>a</sup> | ### | ### | ### | ### | ### |
|---|---|---|---|---|---|
| Pharmacokinetic-evaluable analysis set b | ### (m. m0/) | ### (vvv v0/) | ### (*** **9/) | ### (vvv v·9/) | ### (xx.x%) |
| Immunogenicity analysis set <sup>c</sup> | ### (xx.x%)<br>### (xx.x%) | ### (xx.x%)<br>### (xx.x%) | ### (xx.x%)<br>### (xx.x%) | ### (xx.x%)<br>### (xx.x%) | ### (XX.X%)<br>### (XX.X%) |

<sup>&</sup>lt;sup>a</sup> Safety analysis set includes all subjects who have received at least 1 dose of study agent (JNJ-63723283 or daratumumab, partial or complete) in either safety run-in or Part 2 of the study.

Note: Percentages are calculated with the number of subjects in each group as denominator.

| <b>Display Specifications</b> | |
|-------------------------------|----------|
| Output Identifier | TSIPOP01 |

<sup>&</sup>lt;sup>b</sup> Pharmacokinetic-evaluable analysis set includes all subjects who have received at least 1 dose of daratumumab or JNJ-63723283 and have at least 1 postinfusion sample in either safety run-in or Part 2 of the study.

<sup>&</sup>lt;sup>c</sup> Immunogenicity analysis set include all subjects who have received at least 1 dose of JNJ-63723283 or daratumumab and have appropriate serum samples for detection of antibodies to JNJ-63723283 or daratumumab (i.e., subjects with at least 1 sample obtained after their first dose of JNJ-63723283 or daratumumab) in either safety run-in or Part 2 of the study

TSIDEM-ST01: Summary of Demographics and Baseline Characteristics; Safety Analysis Set (Study 54767414MMY2036)

| Analysis set: Safety | ### | ### | ### | ### | ### |
|---|---|---|---|---|---|
| Age, (years) | | | | | |
| N | ### | ### | ### | ### | ### |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Range | (xx;xx) | (xx;xx) | (xx;xx) | (xx;xx) | (xx;xx) |
| Category, n(%) | | | | | |
| < 65 | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| 65-<75 | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| ≥ 75 | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Sex, n(%) | | | | | |
| N | ### | ### | ### | ### | ### |
| Female | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Male | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Race, n(%) | | | | | |
| N | ### | ### | ### | ### | ### |
| American Indian or Alaska | | | | | |
| Native | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Asian | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Black or African American | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Native Hawaiian or Other Pacific | | | | | |
| Islander | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| White | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Multiple <sup>a</sup> | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Not reported | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Ethnicity, n(%) | | | | | |
| N | ### | ### | ### | ### | ### |
| Hispanic or Latino | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Not Hispanic or Latino | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Not reported | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Weight, kg | | | | | |
| N | ### | ### | ### | ### | ### |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Range | (xx;xx) | (xx;xx) | (xx;xx) | (xx;xx) | (xx;xx) |
| Category, n(%) | | | | | |
| ≤ 65 | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| >65-85 | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| >85 | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Height, cm | | | | | |
| N | ### | ### | ### | ### | ### |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | XX.X | xx.x | xx.x | xx.x |
| Range | (xx;xx) | (xx;xx) | (xx;xx) | (xx;xx) | (xx;xx) |

# TSIDEM-ST01: Summary of Demographics and Baseline Characteristics; Safety Analysis Set (Study 54767414MMY2036)

| Baseline ECOG score, n(%) | | | | | |
|---|---|---|---|---|---|
| N | ### | ### | ### | ### | ### |
| 0 | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| 1 | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| 2 | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |

Key: ECOG=Eastern Cooperative Oncology Group.

Note: Percentages are calculated with the number of subjects in each group with available data as denominator.

#### Programming Notes:

- 1. For sex, race, and ethnicity, categories are presented in alphabetical order.
- 2. For race, each subject must appear in only one category.
- 3. For ordered categories (eg, age (years): <65, >=60), all category levels will be displayed regardless of whether there are zero counts within a level; for categories with no inherent order (eg, race), only category levels with counts >0 will be displayed.

<sup>&</sup>lt;sup>a</sup> If multiple race categories are indicated, the subject's race is include in 'Multiple'.

| TSIDEM02: Summary | of Baseline Disease | Characteristics: Safe | tv Analysis Set ( | Study 54767414MMY2036) |
|---|---|---|---|---|

| • | | <u> </u> | <u>, </u> |
|---|---|---|---|
| Analysis set: Safety | ## | ## | ## |
| Type of myeloma by immunofixation or serum FLC assay, n (%) | | | |
| N | ## | ## | ## |
| IgG | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| IgA | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| IgM | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| IgD | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| IgE | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Light chain | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Kappa | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Lambda | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Biclonal | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Negative Immunofixation | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Not detected | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Type of measurable disease <sup>a</sup> , n(%) | | | |
| N | ## | ## | ## |
| Serum only | | | |
| IgG | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| IgA | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Other b | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Serum and urine | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Urine only | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Serum FLC only | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| NE | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| ISS staging c, n(%) | | | |
| N | ## | ## | ## |
| I | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| II | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| III | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Number of lines of prior therapy <sup>d</sup> | | | |
| N | ## | ## | ## |
| Mean (SD) | ##.# (##.##) | ##.# (##.##) | ##.# (##.##) |
| Median | ## | ## | ## |
| Range | (##; ##) | (##; ##) | (##; ##) |
| Category, n (%) | | | |
| ≤3 | #(XX.X%) | #(XX.X%) | #(XX.X%) |
| > 3 | #(XX.X%) | #(XX.X%) | #(XX.X%) |
| Time from MM diagnosis to first dosing date(years) | | | |
| N | ## | ## | ## |
| Mean (SD) | ##.##(##.###) | ##.##(##.###) | ##.##(##.###) |
| Median | ##.## | ##.## | ##.## |
| Range | (##.#; ##.#) | (##.#; ##.#) | (##.#; ##.#) |

## TSIDEM02: Summary of Baseline Disease Characteristics; Safety Analysis Set (Study 54767414MMY2036)

| Number of lytic bone lesions, n (%) | | | |
|---|---|---|---|
| N | ## | ## | ## |
| None | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| 1-3<br>4-10 | ### (xx.x%)<br>### (xx.x%) | ### (xx.x%)<br>### (xx.x%) | ### (xx.x%)<br>### (xx.x%) |
| More than 10 | ### (XX.X%)<br>### (XX.X%) | ### (XX.X%)<br>### (XX.X%) | ### (XX.X%)<br>### (XX.X%) |
| Presence of diffuse myeloma-related osteopenia, n (%) | | | |
| N | ## | ## | ## |
| Yes | | | |
| No | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| NO | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Number of extramedullary plasmacytomas, n (%) | | | |
| N | ## | ## | ## |
| 0 | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| ≥1 | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Presence of evaluable bone marrow assessment, n (%) | | | |
| N | ## | ## | ## |
| Yes | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| No | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| A/ N | | | |
| % Plasma cells, bone marrow biopsy/aspirate, n (%) | 1111 | 1111 | 1111 |
| N | ## | ## | ## |
| <10 | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| 10-30 | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| >30 | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Cytogenetic risk <sup>e</sup> , n (%) | | | |
| N | ## | ## | ## |
| Standard Risk | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| High Risk <sup>f</sup> | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Del(17p) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| T(4;14) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| T(14;16) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |

## TSIDEM02: Summary of Baseline Disease Characteristics; Safety Analysis Set (Study 54767414MMY2036)

| Baseline ECG | | | |
|---|---|---|---|
| N | ## | ## | ## |
| Normal | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Abnormal, not clinically significant | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Abnormal, clinically significant | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |

Key: ECG = electrocardiogram; FLC = serum free light chain; ISS = International Staging System; MM = multiple myeloma; NE=not evaluable.

Note: Percentages calculated with the number of subjects in each group with available data as denominator.

| <b>Display Specifications</b> | |
|---|---|
| Output Identifier | TSIDEM02 |
| Programming Notes: | |
| 1. No need to show "Not detected" or "NE" categories if no such subjects exist | |

# LSIDEM-ST01: Listing of Demographics and Baseline Characteristics; Safety Analysis set (Study 54767414MMY2036)

| | | | | | | | Baseline | |
|---|---|---|---|---|---|---|---|---|
| | | | | | | | | <u>ECOG</u> |
| <u>Treatment</u> | Site | | Informed | Age (years)/ | | Weight | | <u>Performance</u> |
| Group | ID | Subject ID | Consent Date | Sex/Race | Ethnicity | (kg) | Height (cm) | <u>Score</u> |
| | | | | 30/M | | | | |

Key: ECOG=Eastern Cooperative Oncology Group.

| Display Specifications | |
|---|---|
| Output Identifier | LSIDEM01 |
| Programming Notes: | |
| 1. Sort listing based on treatment group (Safety run-in, Arm A, Arm B), site ID, and subject ID. | |

<sup>&</sup>lt;sup>a</sup> Includes subjects without measurable disease in serum and urine.

<sup>&</sup>lt;sup>b</sup> Includes subjects with IgD, IgM, IgE and biclonal.

 $<sup>^{\</sup>text{c}}$  ISS staging is derived based on the combination of serum  $\beta2\text{-microglobulin}$  and albumin.

<sup>&</sup>lt;sup>d</sup> Based on data recorded on prior systemic therapy eCRF page.

<sup>&</sup>lt;sup>e</sup> Cytogenetic risk is based on FISH or karyotype testing.

f Subject may have more than one high-risk abnormality [del17p, t(4;14) or t(14;16)].

TSIMH01: Summary of Medical History by MedDRA System Organ Class and Preferred term; Safety Analysis Set (Study 54767414MMY2036)

| Analysis set: Safety | ## | ## | ## |
|---|---|---|---|
| Total number of subjects with 1 or more medical history | #(X.X%) | #(X.X%) | #(X.X%) |
| MedDRA system organ class / Preferred term | #(X.X%) | #(X.X%) | #(X.X%) |
| System organ class | #(X.X%) | #(X.X%) | #(X.X%) |
| Preferred term | #(X.X%) | #(X.X%) | #(X.X%) |

Note: Percentages calculated with the number of subjects in each treatment group as denominator. Medical history is coded using MedDRA version 20.X.

| TSIPM01: Summary of Prior Systemic Therapies: Safety Analysis Set (Study 54767414MMY20 | TSIPM01: Summary | of Prior Systemic Tl | herapies: Safety An | alvsis Set (Stud | v 54767414MMY203 |
|---|---|---|---|---|---|
|---|---|---|---|---|---|

| Analysis set: Safety | ## | ## | ## |
|---|---|---|---|
| Total number of subjects with any prior therapies for multiple myeloma, n (%) | #(XX.X%) | #(XX.X%) | #(XX.X%) |
| Prior systemic therapy | #(XX.X%) | #(XX.X%) | # (XX.X%) |
| Prior autologous stem cell transplant (ASCT) | #(XX.X%) | #(XX.X%) | #(XX.X%) |
| Prior radiotherapy | #(XX.X%) | #(XX.X%) | # (XX.X%) |
| Prior cancer-related surgery | #(XX.X%) | #(XX.X%) | #(XX.X%) |
| Prior PI, n (%) | | | |
| Bortezomib | #(XX.X%) | #(XX.X%) | #(XX.X%) |
| Carfilzomib | #(XX.X%) | #(XX.X%) | #(XX.X%) |
| Ixazomib | #(XX.X%) | #(XX.X%) | #(XX.X%) |
| Prior IMiD, n (%) | | | |
| Lenalidomide | #(XX.X%) | #(XX.X%) | #(XX.X%) |
| Pomalidomide | #(XX.X%) | #(XX.X%) | #(XX.X%) |
| Thalidomide | #(XX.X%) | #(XX.X%) | #(XX.X%) |
| Prior PI+IMiD, n (%) | | | |
| Prior corticosteroids, n (%) | | | |
| Dexamethasone | #(XX.X%) | #(XX.X%) | #(XX.X%) |
| Prednisone | #(XX.X%) | #(XX.X%) | #(XX.X%) |
| Prior alkylating agents, n (%) | #(XX.X%) | #(XX.X%) | #(XX.X%) |
| Prior anthracyclines, n (%) | #(XX.X%) | #(XX.X%) | # (XX.X%) |

Note: Percentages calculated with the number of subjects in each group as denominator

### TSICM-ST01: Summary of Concomitant Medications; Safety Analysis Set (Study 54767414MMY2036)

| Analysis set: Safety | ### | ### | ### | ### | ### |
|---|---|---|---|---|---|
| Subjects with one or more concomitant medications | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| ATC Level 2 ATC Level 3 Standardized medication name | ### (xx.x%)<br>### (xx.x%)<br>### (xx.x%) | ### (xx.x%)<br>### (xx.x%)<br>### (xx.x%) | ### (xx.x%)<br>### (xx.x%)<br>### (xx.x%) | ### (xx.x%)<br>### (xx.x%)<br>### (xx.x%) | ### (xx.x%)<br>### (xx.x%)<br>### (xx.x%) |

Note: Percentages calculated with the number of subjects in each group as denominator.

| <b>Display Specifications</b> | |
|-------------------------------|---------|
| Output Identifier | TSICM01 |
| Programming Notes: | |

1. Order by decreasing incidence of ATC level and decreasing incidence of standardized medication name based on the overall total column.

| Display Specifications | |
|------------------------|---------|
| Output Identifier | TSICM02 |
| _ | |

#### Programming note:

- 1. Change the 'concomitant' to 'pre-infusion' in the title and table.
- 2. Order by decreasing incidence of ATC level and decreasing incidence of standardized medication name based on the overall total column.

| <b>Display Specifications</b> | |
|-------------------------------|---------|
| Output Identifier | TSICM03 |

### Programming note:

- 1. Change the 'concomitant' to 'post-infusion' in the title and table.
- 2. Order by decreasing incidence of ATC level and decreasing incidence of standardized medication name based on the overall total column.

| LSICM01: Listing of Pre-infusion | <b>Medications: Safet</b> | v Analysis Set (S | Study 54767414MMY2036) |
|---|---|---|---|

| Treatment Group | Site ID | Subject<br>ID | Visit | Start Date/Time<br>(Study Day) | Medication Coded Term [Verbatim Term] | Dose (unit) | Route |
|---|---|---|---|---|---|---|---|
| Safety run-in | XXX | XXXXXXXX | CYCLE 1 DAY 1 | 2017-11-01T09:00 (1) | CLEMASTINE FUMARATE [TAVEGYL] | 2 (mg) | INTRAVENOUS |
| | | | CYCLE 1 DAY 8 | 2017-11-08T09:00 (8) | CLEMASTINE FUMARATE [TAVEGYL] | 2 (mg) | INTRAVENOUS |
| | | XXXXXXXX | CYCLE 1 DAY 1 | 2017-11-01T09:00 (1) | CLEMASTINE FUMARATE [TAVEGYL] | 2 (mg) | INTRAVENOUS |

Programming note: please sort data by Treatment group (Safety run-in, Arm A, Arm B), site ID, subject ID, start Date/Time

# LSICM02: Listing of Post-infusion Medications; Safety Analysis Set (Study 54767414MMY2036)

| Treatment<br>Group | Site ID | Subject ID | Visit | Start Date<br>(Study Day) | End Date<br>(Study Day) | Medication Coded Term [Verbatim Term] | Dose (unit) | Route | Frequency |
|---|---|---|---|---|---|---|---|---|---|
| Safety run-in | XXX | XXXXXXXX | CYCLE 1 DAY | 2017-11-01 (1) | 2017-11-02 (2) | METHYLPREDNISOLONE [MEDROL] | 20 (mg) | ORAL | Twice Daily |
| | | | CYCLE 1 DAY | 2017-11-08 (8) | 2017-11-08 (9) | METHYLPREDNISOLONE [MEDROL] | 20 (mg) | ORAL | Twice Daily |
| | | XXXXXXXX | CYCLE 1 DAY | 2017-11-01 (1) | 2017-11-02 (2) | METHYLPREDNISOLONE [MEDROL] | 20 (mg) | ORAL | Twice Daily |
| | | XXXXXXXX | CYCLE 1 DAY | 2017-11-01 (1) | 2017-11-02 (2) | METHYLPREDNISOLONE [MEDROL] | 20 (mg) | ORAL | Twice Daily |

Programming note: please sort data by Treatment group (Safety run-in, Arm A, Arm B), site ID, subject ID, Start date.

| LSIPM01: List of Subjects with Prior Cancer-Related Surgery/Procedure; Safety Analysis Set (Study 54767414MMY2036) | | | | | | |
|---|---|---|---|---|---|---|
| Treatment Group | Site<br>ID | Subject ID | Description of Surgery or Procedure | Start Date | End Date | Indication |

# Programming Notes:

1. Listing is sorted by treatment (Safety run-in, Arm A and Arm B), site ID, subject ID, start date of procedure.

| LSIPM02: List | of Prior Radio | therapy; Safety A | nalysis Set (Stud | ly 54767414MMY | 2036) | | |
|---|---|---|---|---|---|---|---|
| Treatment | Site | Subject ID | Start Date | End Date | Location | Indication | Total Dose (Gy) |
| Group | ID | | | | | | |

## Programming Notes:

- 1. Listing is sorted by treatment (Safety run-in, Arm A and Arm B), site ID, subject ID, start date of procedure.
- 2. If indication/location is "Other" and there is a specific description of the indication/location, then the specific description should be displayed

| LSIDEV-ST01: | Listing of S | Subjects with M | Iajor Protocol Deviations; Safety Analysis Set (Study 54767414MMY2036) | |
|---|---|---|---|---|
| Treatment Group | Site ID | Subject ID | Type of Protocol Deviation | Protocol Deviation Verbatim Term |

## Programming Notes:

1. The sort order is Treatment Group (Safety run-in, Arm A and Arm B), Site ID, Subject ID, and Study Day of Deviation.

TSIEX-ST01: Summary of Treatment Cycles, Duration of Study Treatment and Dose Intensity; Safety Analysis Set (Study 54767414MMY2036)

| Analysis set: Safety ### ### Duration of treatment (months) N ### ### Mean (SD) | | | | |
|---|---|---|---|---|
| N ### ### ### Median xx.x (xx.xx) xx.x (xx.xx) xx.x (xx.xx) Number of treatment cycles ### ### ### N ### ### ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) xx.x (xx.xx) Median xx.x xx.x xx.x xx.x Range (xx.xx) (xx.xx) (xx.xx) xx.x ≥ 1 cycle ## (XX.X%) ## (XX.X%) ## (XX.X%) ±# (XX.X%) ## (XX.X%) ±# (XX.X%) *# (XX.XX) ** (XX.XX) ** (XX.X | ### | ### | ### | Analysis set: Safety |
| Mean (SD) xx.x (xx.xx) xx.x (xx.xx) Range (xx,xx) xx.x Number of treatment cycles ### ### N ### ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) Median xx.x (xx.xx) xx.x (xx.xx) Axx.x (xx.xx) xx.x (xx.xx) xx.x (xx.xx) Polycle ## (XX.X%) ## (XX.X%) ≥ 1 cycle ## (XX.X%) ## (XX.X%) ≥ 3 cycles ## (XX.X%) ## (XX.X%) ≥ 4 cycles ## (XX.X%) ## (XX.X%) ≥ 5 cycles ## (XX.X%) ## (XX.X%) Fotal number of daratumumab infusions XXX.X (xX.XXX) XXX.X (xX.XXX) N ### ### ### Mean (SD) XXX.X (XX.XXX) XXX.X (XX.XXX) N ### ### ### Mean (SD) XXX.X (XX.XXX) XXX.X (XX.XXX) N ### ### Median XXX.X (XX.XXX) XXX.X (XX.XXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | Duration of treatment (months) |
| Median Range xx.x x (xx,xx) xx.x (xx,xx) Number of treatment cycles ### ### ### Nean (SD) xx.x (xx.xx) xx.x (xx.xx) Median xx.x (xx.xx) xx.x (xx.xx) Range (xx.xx) (xx.xx) ≥ 1 cycle ## (XX.X%) ## (XX.X%) ≥ 3 cycles ## (XX.X%) ## (XX.X%) ≥ 4 cycles ## (XX.X%) ## (XX.X%) ≥ 5 cycles ## (XX.X%) ## (XX.X%) Fotal number of daratumumab infusions ### (XX.Xxx) ### (XX.Xxx) N Median xx.x (xx.xx) xx.x (xx.xx) Range (xx,xx) (xx,xx) Total dose of daratumumab (mg/kg) ### ### ### N Median xx.x (xx.xx) xx.x (xx.xx) Range (xx,xx) (xx,xx) Dose intensity for daratumumab (mg/kg/cycle) <sup>a</sup> ### ### ### N Median xx.x (xx.xx) xx.x (xx.xx) Relative dose intensity for daratumumab (%) ### ### ### N Median xx.x (xx.xx) xx.x (xx.xx) < | ### | ### | ### | N |
| Range (xx,xx) (xx,xx) Number of treatment cycles ### ### N Mean (SD) xx.x (xx.xx) xx.x (xx.xx) Median xx.x xx.x xx.x Range (xx,xx) (xx,xx) (xx,xx) ≥ 1 cycle ## (XX.X%) ## (XX.X%) ## (XX.X%) ≥ 2 cycles ## (XX.X%) ## (XX.X%) ## (XX.X%) ≥ 3 cycles ## (XX.X%) ## (XX.X%) ## (XX.X%) ≥ 5 cycles ## (XX.X%) ## (XX.X%) ## (XX.X%) Fotal number of daratumumab infusions ### ### ### N ### ### ### Median xx.x xx.x xx.x Range (xx,xx) xx.x xx.x Pose intensity for daratumumab (mg/kg/cycle) and manage ### ### N ### ### Median xx.x xx.x xx.x Relative dose intensity for daratumumab (%) ### ### N ### ### Mean (SD) xx.x xx.x xx.x <tr< td=""><td>xx.x(xx.xx)</td><td>xx.x (xx.xx)</td><td>xx.x(xx.xx)</td><td></td></tr<> | xx.x(xx.xx) | xx.x (xx.xx) | xx.x(xx.xx) | |
| Mean (SD) | XX.X | | XX.X | |
| N ### ### Median xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x <t< td=""><td>(xx;xx)</td><td>(xx;xx)</td><td>(xx;xx)</td><td>Range</td></t<> | (xx;xx) | (xx;xx) | (xx;xx) | Range |
| Mean (SD) xx.x (xx.xx) xx.x (xx.xx) Median xx.x (xx.xx) xx.x (xx.xx) Range (xx;xx) (xx;xx) ≥ 1 cycle ## (XX.X%) ## (XX.X%) ≥ 2 cycles ## (XX.X%) ## (XX.X%) ≥ 3 cycles ## (XX.X%) ## (XX.X%) ≥ 4 cycles ## (XX.X%) ## (XX.X%) ≥ 5 cycles ## (XX.X%) ## (XX.X%) otal number of daratumumab infusions ### ### N ### ### ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) Median xx.x (xx.xx) xx.x (xx.xx) N ### ### ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) N ### ### ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) N ### ### ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) N ### ### ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) N ### ### ### | | | | |
| Median XX.X XX.X Range (XX,XX) (XX,XX) ≥ 1 cycle ## (XX.X%) ## (XX.X%) ≥ 2 cycles ## (XX.X%) ## (XX.X%) ≥ 3 cycles ## (XX.X%) ## (XX.X%) ≥ 4 cycles ## (XX.X%) ## (XX.X%) ≥ 5 cycles ## (XX.X%) ## (XX.X%) Otal number of daratumumab infusions ** ## ## ## ## ## ### Mean (SD) XX.X (XX.XX) XX.X (XX.XX) Median XX.X (XX.XX) XX.X (XX.XX) N ### ## ### ### ### Median XX.X (XX.XX) XX.X (XX.XX) N ### ### ### ### Median XX.X (XX.XX) XX.X (XX.XX) N ### ### ### ### Median XX.X (XX.XX) XX.X (XX.XX) N ### ### ### Mean (SD) XX.X (XX.XX) XX.X (XX.XX) N ### ### ### Median XX.X (XX.XX) XX.X (XX.XX) N ### ### ### Median XX.X (XX.XX) XX.X (XX.XX) | ### | | | |
| Range | xx.x (xx.xx) | | | |
| ≥ 1 cycle | XX.X | | | |
| ≥ 2 cycles | (xx;xx) | | | |
| ≥ 3 cycles | ## (XX.X%) | | ` / | - |
| ≥ 4 cycles ≥ 5 cycles ## (XX.X%) ## (XX.X%) ≥ 5 cycles ## (XX.X%) ## (XX.X%) ## ## ## ## ## ### ### ### Mean (SD) | ## (XX.X%) | | | • |
| ≥ 5 cycles ## (XX.X%) ## (XX.X%) botal number of daratumumab infusions N ### ### Mean (SD) | ## (XX.X%) | | | |
| Mean (SD) | ## (XX.X%) | | | - |
| N ### ### Mean (SD) XX.X (XX.XX) XX.X (XX.XX) Median XX.X XX.X Range (XX;XX) (XX;XX) Stal dose of daratumumab (mg/kg) ### ### Mean (SD) XX.X (XX.XX) XX.X (XX.XX) Median XX.X XX.X Range (XX;XX) XX.X (XX.XX) See intensity for daratumumab (mg/kg/cycle) <sup>a</sup> XX.X XX.X XX.X Mean (SD) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) Median XX.X XX.X XX.X Median XX.X XX.X XX.X Mean (SD) XX.X (XX.XX) XX.X (XX.XX) Median XX.X XX.X XX.X | ## (XX.X%) | ## (XX.X%) | ## (XX.X%) | ≥ 5 cycles |
| Mean (SD) xx.x (xx.xx) xx.x (xx.xx) Median xx.x xx.x Range (xx,xx) (xx,xx) otal dose of daratumumab (mg/kg) ### ### N ### ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) Median xx.x (xx.xx) xx.x (xx.xx) N ### ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) Median xx.x (xx.xx) xx.x (xx.xx) Median xx.x (xx.xx) xx.x (xx.xx) Median xx.x (xx.xx) xx.x (xx.xx) Mean (SD) xx.x (xx.xx) xx.x (xx.xx) Mean (SD) xx.x (xx.xx) xx.x (xx.xx) Mean (SD) xx.x (xx.xx) xx.x (xx.xx) Median xx.x (xx.xx) xx.x (xx.xx) Median xx.x (xx.xx) xx.x (xx.xx) Median xx.x (xx.xx) xx.x (xx.xx) Median xx.x (xx.xx) xx.x (xx.xx) Median xx.x (xx.xx) xx.x (xx.xx) Median <td></td> <td></td> <td></td> <td>otal number of daratumumab infusions</td> | | | | otal number of daratumumab infusions |
| Median Range xx.x (xx;xx) xx.x (xx;xx) Otal dose of daratumumab (mg/kg) ### ### ### N ### ### ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) Median xx.x (xx;xx) (xx;xx) Oose intensity for daratumumab (mg/kg/cycle) and consists of the state of the sta | ### | ### | ### | |
| Range (xx;xx) (xx;xx) Otal dose of daratumumab (mg/kg) ### ### N xx.x (xx.xx) xx.x (xx.xx) Median xx.x xx.x Range (xx;xx) (xx;xx) ose intensity for daratumumab (mg/kg/cycle) and consists of the construction of the c | xx.x(xx.xx) | xx.x (xx.xx) | xx.x(xx.xx) | Mean (SD) |
| Man (SD) | XX.X | XX.X | XX.X | |
| N ### ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) Median xx.x xx.x Range (xx;xx) (xx;xx) Ose intensity for daratumumab (mg/kg/cycle) and serior intensity for daratumumab (mg/kg/cycle | (xx;xx) | (xx;xx) | (xx;xx) | Range |
| Mean (SD) xx.x (xx.xx) xx.x (xx.xx) Median xx.x xx.x Range (xx;xx) (xx;xx) ose intensity for daratumumab (mg/kg/cycle) and serior intensity | | | | otal dose of daratumumab (mg/kg) |
| Median Range xx.x | ### | | | |
| Range (xx;xx) (xx;xx) ose intensity for daratumumab (mg/kg/cycle) <sup>a</sup> ### ### N ### ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) Median xx.x (xx;xx) (xx;xx) Ilative dose intensity for daratumumab (%) ### ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) Median xx.x (xx;xx) (xx;xx) tal number of JNJ-63723283 infusions ### ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) Median xx.x (xx.xx) xx.x (xx.xx) Median xx.x (xx.xx) xx.x (xx.xx) tal dose of JNJ-63723283 (mg) ### ### N ### ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x(xx.xx) | |
| see intensity for daratumumab (mg/kg/cycle) a N | XX.X | XX.X | XX.X | Median |
| N ### ### ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) Median xx.x xx.x Range (xx;xx) (xx;xx) Idative dose intensity for daratumumab (%) ### ### N ### ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) Median xx.x (xx.xx) xx.x (xx.xx) Median xx.x (xx.xx) xx.x (xx.xx) Median xx.x (xx.xx) xx.x (xx.xx) Range (xx;xx) (xx;xx) Ital dose of JNJ-63723283 (mg) ### ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) Mean (SD) xx.x (xx.xx) xx.x (xx.xx) | (xx;xx) | (xx;xx) | (xx;xx) | Range |
| Mean (SD) xx.x (xx.xx) xx.x (xx.xx) Median xx.x xx.x Range (xx;xx) (xx;xx) Elative dose intensity for daratumumab (%) ### ### N ### ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) Median xx.x (xx,xx) (xx;xx) Mean (SD) xx.x (xx.xx) xx.x (xx.xx) Median xx.x (xx.xx) xx.x (xx.xx) Median xx.x (xx.xx) (xx;xx) Median xx.x (xx.xx) (xx;xx) Metal dose of JNJ-63723283 (mg) ### ### N ### ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) | | | | ose intensity for daratumumab (mg/kg/cycle |
| Median Range xx.x (xx;xx) xx.x (xx;xx) elative dose intensity for daratumumab (%) ### ### ### ### N ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) Median xx.x xxx xx.x (xx.xx) xx.x (xx.xx) Otal number of JNJ-63723283 infusions ### ### ### ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) Median xx.x xxx xx.x (xx.xx) xx.x (xx.xx) Median xx.x (xx.xx) xx.x (xx.xx) xx.x (xx.xx) Otal dose of JNJ-63723283 (mg) ### ### ### N ### ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) | ### | | | |
| Range (xx;xx) (xx;xx) elative dose intensity for daratumumab (%) ### ### N ### ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) Median xx.x (xx.xx) (xx;xx) Otal number of JNJ-63723283 infusions ### ### N ### ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) Median xx.x (xx.xx) (xx;xx) Otal dose of JNJ-63723283 (mg) ### ### N ### ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) | xx.x(xx.xx) | |
| Mean (SD) | XX.X | XX.X | XX.X | |
| N ### ### ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) Median xx.x xx.x Range (xx;xx) (xx;xx) tal number of JNJ-63723283 infusions ### ### N ### ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) Median xx.x xx.x Range (xx;xx) (xx;xx) tal dose of JNJ-63723283 (mg) ### ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) | (xx;xx) | (xx;xx) | (xx;xx) | Range |
| Mean (SD) xx.x (xx.xx) xx.x (xx.xx) Median xx.x xx.x Range (xx;xx) (xx;xx) Otal number of JNJ-63723283 infusions ### ### N ### ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) Median xx.x xx.x Range (xx;xx) (xx;xx) Otal dose of JNJ-63723283 (mg) ### ### N ### ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) | | | | elative dose intensity for daratumumab (%) |
| Median xx.x xx.x Range (xx;xx) (xx;xx) Stal number of JNJ-63723283 infusions ### ### ### N ### ### ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) Median xx.x xx.x Range (xx;xx) (xx;xx) Otal dose of JNJ-63723283 (mg) ### ### ### N ### ## ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) | ### | ### | ### | N |
| Median xx.x xx.x Range (xx;xx) (xx;xx) Stal number of JNJ-63723283 infusions ### ### N ### ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) Median xx.x xx.x Range (xx;xx) (xx;xx) Stal dose of JNJ-63723283 (mg) ### ### N ### ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | Mean (SD) |
| Range (xx;xx) (xx;xx) stal number of JNJ-63723283 infusions ### ### N ### ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) Median xx.x xx.x Range (xx;xx) (xx;xx) stal dose of JNJ-63723283 (mg) ### ### N ### ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) | XX.X | | | |
| Mean (SD) | (xx;xx) | | | |
| N ### ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) Median xx.x xx.x Range (xx;xx) (xx;xx) otal dose of JNJ-63723283 (mg) ### ### N ### ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) | | | | otal number of INI-63723283 infusions |
| Mean (SD) xx.x (xx.xx) xx.x (xx.xx) Median xx.x xx.x Range (xx;xx) (xx;xx) otal dose of JNJ-63723283 (mg) ### ### N ### ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) | ### | ### | ### | |
| Median xx.x xx.x Range (xx;xx) (xx;xx) stal dose of JNJ-63723283 (mg) ### ### N ### ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) | | | | |
| Range (xx;xx) (xx;xx) otal dose of JNJ-63723283 (mg) N ### ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) | XX.X (XX.XX) | | | |
| tal dose of JNJ-63723283 (mg) N ### ### Mean (SD) | XX.X | | | |
| N ### ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) | (xx;xx) | (xx;xx) | (xx;xx) | Range |
| N ### ### Mean (SD) xx.x (xx.xx) xx.x (xx.xx) | | | | otal dose of JNJ-63723283 (mg) |
| Mean (SD) xx.x (xx.xx) xx.x (xx.xx) | ### | ### | ### | |
| | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | XX.X | XX.X | XX.X | Median |
| Range (xx;xx) (xx;xx) | (xx;xx) | | | |

TSIEX-ST01: Summary of Treatment Cycles, Duration of Study Treatment and Dose Intensity; Safety Analysis Set (Study 54767414MMY2036)

| Dose intensity for JNJ-63723283 (mg/cycle) b | | | |
|---|---|---|---|
| N | ### | ### | ### |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Range | (xx;xx) | (xx;xx) | (xx;xx) |
| Relative dose intensity for JNJ-63723283 (%) | | | |
| N | ### | ### | ### |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Range | (xx;xx) | (xx;xx) | (xx;xx) |

<sup>&</sup>lt;sup>a</sup> Dose intensity (mg/kg/cycle) is calculated as the sum of total doses (mg/kg) received in all cycles divided by the number of treatment cycles on daratumumab.

Note: The relative dose intensity (%) is the ratio of total actually received dose and total planned dose.

TSIEXP02: Summary of Treatment Cycle Delays, Incidences of and Reasons for Study Treatment Dose Modifications; Safety Analysis Set (Study 54767414MMY2036)

| Analysis set: Safety | ## | ## |
|----------------------------|------------|------------|
| Subjects with cycle delays | ## (XX.X%) | ## (XX.X%) |
| Reason for cycle delays | | |
| Adverse event | ## (XX.X%) | ## (XX.X%) |
| Other | ## (XX.X%) | ## (XX.X%) |
| Subjects with dose delays | | |
| Daratumumab | ## (XX.X%) | ## (XX.X%) |
| Reason for delays | | |
| Adverse event | ## (XX.X%) | ## (XX.X%) |
| Other | ## (XX.X%) | ## (XX.X%) |
| JNJ-63723283 | ## (XX.X%) | ## (XX.X%) |
| Reason for delays | | |
| Adverse event | ## (XX.X%) | ## (XX.X%) |
| Other | ## (XX.X%) | ## (XX.X%) |
| Subjects with dose skipped | | |
| Daratumumab | ## (XX.X%) | ## (XX.X%) |
| Reason for skipping | | |
| Adverse event | ## (XX.X%) | ## (XX.X%) |
| Other | ## (XX.X%) | ## (XX.X%) |

<sup>&</sup>lt;sup>b</sup> Dose intensity (mg/cycle) is calculated as the sum of total doses (mg) received in all cycles divided by the number of treatment cycles on JNJ-63723283.

| TSIEXP02: Summary of Treatment Cycle Delays, Incidences of and Reasons for Study Treatment |
|---|
| Dose Modifications; Safety Analysis Set (Study 54767414MMY2036) |

| JNJ-63723283 | ## (XX.X%) | ## (XX.X%) |
|---------------------|------------|------------|
| Reason for skipping | | |
| Adverse event | ## (XX.X%) | ## (XX.X%) |
| Other | ## (XX.X%) | ## (XX.X%) |

Note: Percentages calculated with the number of subjects in each group as denominator.

# TSIEXP03: Summary of Action Taken During the Infusion; Safety Analysis Set (Study 54767414MMY2036)

| Analysis set: Safety | ## | ## |
|---------------------------------------|------------|------------|
| Subjects with infusion interrupted | | |
| Daratumumab | ## (XX.X%) | ## (XX.X%) |
| Reason for infusion interrupted | | |
| Adverse event | ## (XX.X%) | ## (XX.X%) |
| Other | ## (XX.X%) | ## (XX.X%) |
| JNJ-63723283 | ## (XX.X%) | ## (XX.X%) |
| Reason for infusion interrupted | | |
| Adverse event | ## (XX.X%) | ## (XX.X%) |
| Other | ## (XX.X%) | ## (XX.X%) |
| Subjects with infusion rate decreased | | |
| Daratumumab | ## (XX.X%) | ## (XX.X%) |
| Reason for infusion rate decreased | | |
| Adverse event | ## (XX.X%) | ## (XX.X%) |
| Other | ## (XX.X%) | ## (XX.X%) |
| JNJ-63723283 | ## (XX.X%) | ## (XX.X%) |
| Reason for infusion rate decreased | | |
| Adverse event | ## (XX.X%) | ## (XX.X%) |
| Other | ## (XX.X%) | ## (XX.X%) |
| Subjects with infusion aborted | | |
| Daratumumab | ## (XX.X%) | ## (XX.X%) |
| Reason for infusion aborted | | |
| Adverse event | ## (XX.X%) | ## (XX.X%) |
| Other | ## (XX.X%) | ## (XX.X%) |
| JNJ-63723283 | ## (XX.X%) | ## (XX.X%) |
| Reason for infusion aborted | | |
| Adverse event | ## (XX.X%) | ## (XX.X%) |
| Other | ## (XX.X%) | ## (XX.X%) |

Note: Percentages calculated with the number of subjects in each group as denominator.

### LSIEX-ST01: Listing of Treatment Exposure; Safety Analysis Set (Study 54767414MMY2036)

| | | | | | | | | | | | Reason for | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | Infusion | | | | Reason for | | Action | |
| | | | | | Date | Total | | Action Planned | Action Planned | Action Taken | Taken | <u>If 'INFUSION</u> |
| Treatment | Site | Subject | Study | | (Study | Dose | Start/End | Prior to Infusion | Prior to | <u>During</u> | <b>During</b> | INTERRUPTED', Interruption |
| <u>Group</u> | <u>ID</u> | ID | Drug | Visit | Day) | (mg) | <u>Time</u> | <u>Start</u> | Infusion Start | <u>Infusioin</u> | <u>Infusion</u> | Start/End Time |

### Programming Notes:

The sort order is Treatment Group (Safety run-in, Arm A, Arm B), Site ID, Subject ID, Study Drug and Infusion Date

### LEFRSP01: Listing of Efficacy Variable Based on Investigator Assessment; Safety Analysis Set (Study 54767414MMY2036)

| | | | | | | | | | Date of Last | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatm | | | | | Date of Best Resp. | Date of | | Reason | Disease | | Date of Death/ | |
| ent | | Subject | Measurable | Best | (Study Day) | PD | Reason | for PD | Assessment | PFS | Last Date Known to be | OS |
| Group | Site ID | ID | Disease Type | Resp. | | (Study Day) | for PD | Censoring | (Study Day) | (Month) | Alive (Study Day) | (Month) |
| Arm A | XX | XX | Serum | CR | 2018-06-04 (XX) | | | XX | 2018-06-14 (xx) | 2.4+ | 2018-06-14 (xx) | 2.4+ |

Key: sCR=stringent complete response; CR=complete response; VGPR=very good partial response; PR=partial response; MR=minimal response; SD=stable disease; PD=progression disease; NE=not evaluable. Key: OS=Overall Survival; PFS=Progression-free Survival; Resp.=Response. +: Censoring.

## Programming notes:

Sort the listing by Treatment group (Arm A, Arm B), Site ID, and Subject ID.

TSFAE-ST01: Overview of Treatment-emergent Adverse Events; Safety Analysis Set (Study 54767414MMY2036)

| Analysis set: Safety | ### | ### | ### | ### |
|---|---|---|---|---|
| Any TEAE | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| At least one related <sup>a</sup> | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| At least one related to daratumumab | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| At least one related to JNJ-63723283<br>Maximum toxicity grade | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Grade 1 | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Grade 2 | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Grade 3 | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Grade 4 | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Grade 5 | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Any serious TEAE | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| At least one related <sup>a</sup> | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| At least one related to daratumumab | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| At least one related to JNJ-63723283 | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| TEAE leading to discontinuation of study treatment <sup>b</sup> | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| TEAE leading to discontinuation of | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| daratumumab | , | , | , | ` , |
| At least one related to daratumumab | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| TEAE leading to discontinuation of JNJ-63723283 | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| At least one related to JNJ-63723283 | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| TEAE with outcome of death | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| At least one related to daratumumab | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| At least one related to JNJ-63723283 | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |

Key: TEAE = treatment-emergent adverse event.

<sup>&</sup>lt;sup>b</sup> Includes those subjects indicated as having discontinued treatment due to an adverse event on the end of treatment CRF page. Note: Adverse events are coded using MedDRA version XX.X. Percentages are calculated with the number of subjects in each group as denominator.

| Display Specifications | |
|------------------------|--------|
| Output Identifier | TSFAE0 |

Programming Notes:

- 1. TEAE with outcome of death are based on an AE outcome equal to Fatal or toxicity grade of 5 from AE page.
- 2. An AE is considered to result in discontinuation of study agent if the "action taken regarding study agent" is "drug withdrawn" on the AE eCRF page. If an attribute of the AE is missing, it will not be imputed.
- 3. An AE is considered to result in discontinuation of study treatment if the reason for termination on the End of Treatment disposition page is AE.

<sup>&</sup>lt;sup>a</sup> TEAEs related to at least 1 of the 2 study treatments: daratumumab and JNJ-63723283.

TSFAE-ST02: Treatment-emergent Adverse Events by System Organ Class and Preferred Term; Safety Analysis Set (Study 54767414MMY2036)

| Analysis set: Safety | ### | ### | ### | ### |
|---|---|---|---|---|
| Total number of subjects with TEAE<br>MedDRA system organ<br>class/preferred term | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| System organ class<br>Preferred term | ### (xx.x%)<br>### (xx.x%) | ### (xx.x%)<br>### (xx.x%) | ### (xx.x%)<br>### (xx.x%) | ### (xx.x%)<br>### (xx.x%) |
| System organ class<br>Preferred term | ### (xx.x%)<br>### (xx.x%) | ### (xx.x%)<br>### (xx.x%) | ### (xx.x%)<br>### (xx.x%) | ### (xx.x%)<br>### (xx.x%) |

Key: TEAE = treatment-emergent adverse event,

Note: Subjects are counted only once for any given event, regardless of the number of times they actually experienced the event. Adverse events are coded using MedDRA Version XX.X. Percentages are calculated with the number of subjects in each group as denominator.

| <b>Display Specifications</b> | |
|-------------------------------|---------|
| Output Identifier | TSFAE02 |
| Programming Notes: | |

Programming Notes:

1. For any uncoded system organ class, present system organ class in table as "Uncoded"; for any uncoded preferred terms, present 'Uncoded' and add verbatim in parenthese next to the preferred term.

## LSFAE01: Listing of Treatment-emergent Adverse Events; Safety Analysis set (Study 54767414MMY2036)

| Treatment<br>Group | Site<br>ID | Subject<br>ID | Onset Date<br>(Study Day) | End Date<br>(Study Day) | Preferred<br>Term | SAE? | | | Relationship to <sup>a</sup> | | lationship to <sup>a</sup> Action Taken with <sup>b</sup> | | IRR Associated with <sup>c</sup> | | Immune<br>Mediated?<br>(Y/N) | A DLT ?<br>(Y/N) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | - | Dara | JNJ-283 | Dara | JNJ-283 | <del>-</del> | Dara | JNJ-283 | | |
| xxx | XXX | XXX | 2014-06-21 (1) | 2014-06-21 (1) | Cough | No | 1 | VL | NR | DI | DNC | RECOVERED/<br>RESOLVED | Y | N | N | N |
| | | | 2014-06-29 (9) | 2014-06-30<br>(10) | Blood<br>blister | Yes | 3 | NR | VL | DI | DW | RECOVERED/<br>RESOLVED | N | N | N | Y |

Key: Dara=daratumumab. JNJ-283=JNJ-63723283. SAE = Serious adverse event. IRR=infusion related reaction. DLT=dose-limiting toxicity.

Note: Adverse events are coded using MedDRA version XX.X.

| Display Specifications | |
|------------------------|---------|
| Output Identifier | LSFAE01 |

Programming notes:

1. Sort the list by treatment group (Safety run-in, Arm A, Arm B), site ID, subject ID, Onset Date

| <b>Display Specifications</b> | |
|-------------------------------|---------|
| Output Identifier | LSFAE02 |

Programming notes:

- 1. Update 'Treatment-emergent Adverse Events' in the title to 'Treatment-emergent Serious Adverse Events'.
- 2. Remove the 'SAE?' column
- 3. Delete the 'SAE=Serious adverse event' in the footnote.
- 4. Sort the list by treatment group (Safety run-in, Arm A, Arm B), site ID, subject ID, Onset Date

<sup>&</sup>lt;sup>a</sup>: NR = Not Related. DO = Doubtful, Poss. = Possible, Prob. = Probable, VL = Very Likely.

b: DI = Drug Interrupted, DNC = Dose Not Changed, DR = Dose Reduced, DW = Drug Withdrawn, NA = Not Applicable, UN = Unknown.

<sup>&</sup>lt;sup>c</sup>: Y=Yes. N=No. NA=Not Applicable. UN=Unknown.

**Display Specifications** 

Output Identifier LSFAE03

Programming notes:

- 1. Update 'Treatment-emergent Adverse Events' in the title to 'Treatment-emergent Grade 3 or 4 Adverse Events'.
- 2. Sort the list by treatment group (Safety run-in, Arm A, Arm B), site ID, subject ID, Onset Date

### **Display Specifications**

Output Identifier LSFAE04

Programming notes:

- 1. Update 'Treatment-emergent Adverse Events' in the title to 'Subjects who Discontinued All Study Treatment Because of 1 or More Treatment-emergent Adverse Events'.
- 2. Sort the list by treatment group (Safety run-in, Arm A, Arm B), site ID, subject ID, Onset Date

### **Display Specifications**

Output Identifier LSFAE05

Programming notes:

- 1. Update 'Treatment-emergent Adverse Events' in the title to 'Subjects who Discontinued Any Study Drugs Because of 1 or More Treatment-emergent Adverse Events'.
- 2. Sort the list by treatment group (Safety run-in, Arm A, Arm B), site ID, subject ID, Onset Date

### **Display Specifications**

Output Identifier LSFAE06

Programming notes:

- 1. Update 'Treatment-emergent Adverse Events' in the title to 'Infusion Related Reactions'.
- 2. Sort the list by treatment group (Safety run-in, Arm A, Arm B), site ID, subject ID, Onset Date
| Display | Cn. | agifia | ations |
|---------|-----------|--------|--------|
| Dispiay | $o_{\mu}$ | CUIIC | auvus |

Output Identifier LSFAE07

Programming notes:

- 1. Update 'Treatment-emergent Adverse Events' in the title to 'Immune Mediated Adverse Events'.
- 2. Remove the 'Immune Mediated? (Y/N)' column.
- 3. Sort the list by treatment group (Safety run-in, Arm A, Arm B), site ID, subject ID, Onset Date

### **Display Specifications**

Output Identifier LSFAE08

Programming notes:

- 1. Update 'Treatment-emergent Adverse Events' in the title to 'Treatment-emergent Adverse Events Leading to Cycle Delay or Dose Modifications'.
- 2. Sort the list by treatment group (Safety run-in, Arm A, Arm B), site ID, subject ID, Onset Date

### **Display Specifications**

Output Identifier LSFAE09

- 1. Update 'Treatment-emergent Adverse Events 'Treatment-emergent Adverse Events Leading to Infusion Interrupted, Infusion Rate Decreased or Infusion Aborted'.
- 2. Sort the list by treatment group (Safety run-in, Arm A, Arm B), site ID, subject ID, Onset Date

### LSFAE10: Listing of Subjects Who Had New Malignancies; Safety Analysis set (Study 54767414MMY2036)

| Treatment<br>Group | Site ID | Subject<br>ID | Line<br>Number | Diagnosis | Diagnosis<br>Date (Study<br>Day) | Existing malignancy<br>(Y/N) / Initiation<br>Diagnosis Date if 'Y'<br>(Study Day) | pathology (Y/N) / | | | Total No./Dose<br>(mg)of JNJ-283<br>Infusions | | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxx | XXX | XX | 1 | ACUTE<br>MONOBLASTI<br>C LEUKEMIA | | Y/2005-05-01 (-100) | Y/Biopsy | III/ISS | 15/300 | 10/2400 | Curative<br>Surgery | RECOVERED/R<br>ESOLVED |

Key: Dara= daratumumab. JNJ-283=JNJ-63723283.

### LSFDTH-ST01: Listing of Subjects Who Died During the Study; Safety Analysis Set (Study 54767414MMY2036)

| | | | | Total No. of JNJ-283 | | Primary Cause of | Relatio | nship to <sup>a</sup> |
|---|---|---|---|---|---|---|---|---|
| | | | Total No. of Dara | Infusions/Total Dose | | Death | | |
| | | | Infusions/Total Dose (mg/kg) | (mg)/Study Day of Last | Date of Death | (If 'AE', Preferred | | |
| Treatment Group | Site ID | Subject ID | /Study Day of Last Infusion | <u>Infusion</u> | (Study Day) | Term) | Dara | JNJ-283 |
| Infliximab 5 mg/kg | XX | SSSS-PPPP | 20/320/270 | 8/1920/270 | 2017-07-21 (xx) | AE(Upper | NR | NR |
| | | | | | | respiratory tract | | |
| | | | | | | infection) | | |

Key: Dara=daratumumab. JNJ-283=JNJ-63723283

Note: Adverse events are coded using MedDRA version XX.X.

| Display Specifications | | |
|------------------------|-------------------|----------|
| | Output Identifier | LSFDTH01 |

Programming Notes:

1. Sort listing based on treatment group (Safety run-in, Arm A, Arm B), site ID, subject ID.

38

<sup>&</sup>lt;sup>a</sup>: NR = Not Related. DO = Doubtful, Poss. = Possible, Prob. = Probable, VL = Very Likely.

| TSFLAB-ST07: Shift Table of Baseline versus Worst | Toxicity Grade during Treatment in Hematological Test; Safety Analysis Set (Study |
|---|---|
| 54767414MMY2036) | |

| | | - | Treatment Gro | up and Evaluation at | baseline | |
|---|---|---|---|---|---|---|
| | N | Grade 0 | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Analysis set: Safety | ### | | | | | |
| WBC low (Leukopenia) | | | | | | |
| Post-baseline | ### | | | | | |
| Grade 0 | | ## | ## | ## | ## | ## |
| Grade 1 | | ## | ## | ## | ## | ## |
| Grade 2 | | ## | ## | ## | ## | ## |
| Grade 3 | | ## | ## | ## | ## | ## |
| Grade 4 | | ## | ## | ## | ## | ## |

Note: N is the number of subjects with non-missing values for the specific lab test at baseline and at least one postbaseline visit during treatment. The laboratory toxicity grades are derived based on the NCI CTCAE (National Cancer Institute Common Terminology Criteria for Adverse Events) Version 4.03.

| <b>Display Specifications</b> | |
|-------------------------------|----------|
| Output Identifier | TSFLAB01 |
| Programming Notes: | |

1. Parameters: Platelets low (Thrombocytopenia), Neutrophils low (Neutropenia), Hemoglobin low (Anemia), and Lymphocytes low (Lymphocytopenia)

| Display Specifications | |
|------------------------|----------|
| Output Identifier | TSFLAB02 |

- 1. Update 'Hematology' in the title to 'Chemistry'
- 2. List for parameters: ALT high, AST high, Creatinine high, Sodium high (Hypernatremia), Sodium low (Hyponatremia), Potassium high (Hyperkalemia), Potassium low (Hypokalemia), Bilirubin high (hyperbilirubinemia), Alkaline phosphatase high, Corrected calcium high (Hypercalcemia), Corrected calcium low (Hypocalcemia), amylase high (hyperamylasemia), total lipase high (hyperlipasemia)

### LSFLAB-ST01: Listing of Hematology Laboratory Values; Safety Analysis Set (Study 54767414MMY2036)

Treatment Group

Site ID

Subject ID

Parameter (Unit)

Visit

Assessment Date (Study Day)

Result xx

Normal Range xx-xx

### **Display Specifications**

Output Identifier LSFLAB01

Programming Notes:

- 1. Update 'Hematology' in the title to 'Other'
- 2. List for parameters: Thyroid Stimulating Hormone; Free triiodothyronine (T3); Total triiodothyronine (T3); Free thyroxine (T4)
- 3. Unscheduled results or multiple results taken at the same visit will be reported here.
- 4. The standard sort order is Treatment Group, Site ID, Subject ID, Parameter, and Assessment Date.

### **Display Specifications**

Output Identifier LSFVS01

- 1. Update 'Hematology' in the title to 'Vital Signs'
- 2. List for parameters: Diastolic blood pressure (mmHg), Systolic blood pressure (mmHg) and weight (kg)
- 3. Unscheduled results or multiple results taken at the same visit will be reported here.
- 4. The standard sort order is Treatment Group, Site ID, Subject ID, Parameter, and Assessment Date.
- 5. Remove the 'Normal Range' column.

| LSFECG-ST01: Listin | ng of ECG Results: | ; Safety Anal | ysis Set (Stud | y 54767414MMY2036) |
|---|---|---|---|---|
| ESTECO STOTT EISTE | -5 or | , ~ | , 525 200 (200 | , |

Treatment Group







Assessment Date (Study Day)

Oerall Interpretation

If 'Abnormal', Clinically Significant? (Y/N)

# **Display Specifications**

Output Identifier

LSFECG01

- 1. Unscheduled results or multiple results taken at the same visit will be reported here.
- 2. The standard sort order is Treatment Group, Site ID, Subject ID, Parameter, and Assessment Date.

TPK-ST07: Summary of Daratumumab Concentrations (ug/mL); Pharmacokinetic-evaluable Analysis Set (Study 54767414MMY2036)

| Analysis set: pharmacokinetic-evaluable | | | | |
|---|---|---|---|---|
| analysis set | ## | ## | ## | ## |
| Cycle 1 Day 1 | | | | |
| N | ### | ### | ### | ### |
| Mean (SD) | x.xx (x.xxx) | x.xx (x.xxx) | x.xx (x.xxx) | x.xx (x.xxx) |
| Median | XXX.X | XXX.X | XXX.X | xxx.x |
| Range | (xxx.x, xxx.x) | (xxx.x, xxx.x) | (xxx.x, xxx.x) | (xxx.x, xxx.x) |
| CV (%) | XXX | XXX | XXX | xxx |
| Geometric mean | X.XX | X.XX | X.XX | X.XX |
| Cycle 2 Day 1 | | | | |
| N | ### | ### | ### | ### |
| Mean (SD) | x.xx (x.xxx) | x.xx (x.xxx) | x.xx (x.xxx) | x.xx (x.xxx) |
| Median | XXX.X | XXX.X | XXX.X | xxx.x |
| Range | (xxx.x, xxx.x) | (xxx.x, xxx.x) | (xxx.x, xxx.x) | (xxx.x, xxx.x) |
| CV (%) | XXX | XXX | XXX | xxx |
| Geometric mean | x.xx | X.XX | X.XX | X.XX |
| Cycle 3 Day 1 | | | | |
| N | ### | ### | ### | ### |
| Mean (SD) | x.xx (x.xxx) | x.xx (x.xxx) | x.xx (x.xxx) | x.xx (x.xxx) |
| Median | XXX.X | XXX.X | XXX.X | XXX.X |
| Range | (xxx.x, xxx.x) | (xxx.x, xxx.x) | (xxx.x, xxx.x) | (xxx.x, xxx.x) |
| CV (%) | XXX | XXX | XXX | XXX |
| Geometric mean | X.XX | X.XX | X.XX | X.XX |

Key: SD = standard deviation, CV = coefficient of variation.

Note: Table includes subjects who received at least 1 administration of daratumumab and have at least 1 pharmacokinetic sample concentration value after the first infusion.

Note: Predose samples with a time of collection prior to the start of infusion for Cycle 1 Day 1, and up to 6 hours prior to the start of infusion for other predose samples will be included from summary statistics. Postdose samples with a time of collection before the end of infusion or more than 15 min after the end of infusion will be excluded from summary statistics.

| <b>Display Specifications</b> | |
|-------------------------------|-----------|
| Output Identifier | TPKCONC01 |
| Programming notes: | |

- 1. Present all available visits.
- 2. For visits of '4 weeks after last dose' and '8 weeks after last dose', data are displayed in the postinfusion column.

| <b>Display Specifications</b> | |
|-------------------------------|-----------|
| Output Identifier | TPKCONC02 |

- 1. Change 'Daratumumab' in the title to 'JNJ-63723283'.
- 2. Present all available visits.
- 3. For visits of '4 weeks after last dose' and '8 weeks after last dose', data are displayed in the postinfusion column.





Note: At each time point, concentration values are plotted on linear scale, and the error bars are mean +/- standard deviation.

Note: Predose samples with a time of collection before the start of infusion for Cycle 1 Day 1, and up to 6 hours prior to the start of infusion for other predose samples will be included from summary statistics. Postdose samples with a time of collection before the end of infusion or more than 15 min after the end of infusion will be excluded from summary statistics.

| Display Specifications | |
|------------------------|-----------|
| Output Identifier | GPKCONC01 |
| D ' 11 ' | |

- 1. Present all available visits in x-axis.
- 2.

| <b>Display Specifications</b> | |
|-------------------------------|-----------|
| Output Identifier | GPKCONC02 |
| Programming Notes: | |

- 1. Change 'Daratumumab' in the title to 'JNJ-63723283'
- 2. Present all available visits in x-axis.

# TPKIR-ST01: Summary of Anti-daratumumab Antibodies Status; Immunogenicity Analysis Set (Study 54767414MMY2036)

| Analysis set: immunogenicity | ### | ### | ### |
|---|---|---|---|
| Subjects with appropriate samples <sup>a</sup> | ### | ### | ### |
| Subjects with baseline positive samples <sup>b,c</sup> | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Subjects positive for anti-daratumumab antibodies <sup>b,d</sup> | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Peak titer | 11111 | 11111 | 11111 |
| 1:20 | ### | ### | ### |
| Subjects positive for neutralizing | | | |
| antibodies | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| Subjects negative for anti-daratumumab antibodies <sup>b,e</sup> | ### (xx.x%) | ### (xx.x%) | ### (xx.x%) |
| antibodies Subjects negative for anti-daratumumab | | , | , |

<sup>&</sup>lt;sup>a</sup> Subjects with appropriate samples had 1 or more samples obtained after their first daratumumab administration.

### **Display Specifications**

Output Identifier TPKIR01

Programming notes:

- 1. Please remove row of "Peak titer" if there is no subject positive for antibodies to daratumumab.
- 2. Please remove 'd' if there are no subject positive for antibody to daratumumab, and change the label 'e' to 'd'.

### **Display Specifications**

Output Identifier TPKIR02

- 1. Change 'Daratumumab' to 'JNJ-63723283' in the whole table.
- 2. Please remove row of "Peak titer" if there is no subject positive for antibodies to JNJ-63723283.
- 3. Please remove 'd' if there are no subject positive for antibody to JNJ-63723283, and change the label 'e' to 'd'.

<sup>&</sup>lt;sup>b</sup> Denominator is subjects with appropriate samples.

<sup>&</sup>lt;sup>c</sup> Subjects with baseline samples positive had samples positive for anti-daratumumab antibodies at baseline, regardless of status after first daratumumab administration.

<sup>&</sup>lt;sup>d</sup> Subjects positive for anti-daratumumab antibodies includes all subjects who were positive (treatment-boosted or treatment-induced) at any time after their first daratumumab administration. Subjects with baseline positive samples and without increased titer after treatment are not considered treatment-boosted.

<sup>&</sup>lt;sup>e</sup> Excludes subjects who were positive at any time.

| LPKIR-ST01: | List of Sub | jects Positive fo | r Anti-daratum | umab Antibodies | Status; Immun | e Response-evaluab | le Analysis Set (Study 54 | 767414MMY2036) |
|---|---|---|---|---|---|---|---|---|
| | | | | Infusion Related | | Toxicity | Daratumumab | Antibody to |
| Treatment Group | Subject ID | Visit/Time Point | Infusion Given? | Reaction | Serious | Grade | Conc. (µg/mL) | Daratumumab Titer |
| | | CYCLE 1 DAY | | | | | | |
| Safety run-in | ###### | 1/PREDOSE | Yes | Yes | No | 1 | LLOQ | NEGTIVE |
| | | CYCLE 2 DAY | | | | | | |
| | | 1/PREDOSE | No | NA | | | 443.7 | 1:20 |

Key: NA= not applicable.

| Display Specifications | |
|------------------------|-----------|
| Output Identifier | LPKCONC01 |
| D : 31 / | |

Programming Notes:

- 1. Listing sort: Treatment Group, Subject ID, and Visit.
- 2. This listing should include all visits where PK sampling was performed for subjects positive for ADA. The titer column will either present the actual titer value (which means they were positive), will be 'NEGATIVE' if there is no titer value (which means they were negative at that visit), or will be "NA" if there was no titer sample at that visit.

| <b>Display Specifications</b> | |
|---------------------------------------|-----------|
| Output Identifier | LPKCONC02 |
| · | |

- 1. Change the 'daratumumab' to 'JNJ-63723283' in the listing.
- 2. Listing sort: Treatment Group, Subject ID, and Visit.
- 3. This listing should include all visits where PK sampling was performed for subjects positive for ADA. The titer column will either present the actual titer value (which means they were positive), will be 'NEGATIVE' if there is no titer value (which means they were negative at that visit), or will be "NA" if there was no titer sample at that visit.



GBMK01: Plot of Percent of Total Natural Killer Cells in Blood Over Time; Safety Analysis Set (Study 54767414MMY2036)

- 1. Display the treatment groups as 'Safety Run-in' or 'Arm A',
- 2. Display the scheduled visits for this study.
- 3. Update the y-lab as appropriate.

| · | | | | | • | - | • | • | ly 54767414MMY2036) Change from Baseline | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | N | Mean | SD | Med | Min | Max | Base<br>Mean | N | Mean | SD | Med | Min | Max |
| Percent of total natural killer cells (%) Safety Run-in | | | | | | | | | | | | | |
| Baseline | XXX | XXX.XX | XXX.XXX | XXX.XX | XX.X | XXX.X | XXX.XX | | | | | | |
| Cycle 1 Day 8 | XXX | XXX.XX | XXX.XXX | XXX.XX | XX.X | XXX.X | XXX.XX | XXX | XXX.XX | XXX.XXX | XXX.XX | XX.X | XXX.X |
| Cycle 1 Day 15 | XXX | XXX.XX | XXX.XXX | XXX.XX | XX.X | XXX.X | XXX.XX | XXX | XXX.XX | XXX.XXX | XXX.XX | XX.X | XXX.X |
| | XXX | XXX.XX | XXX.XXX | XXX.XX | XX.X | XXX.X | XXX.XX | XXX | XXX.XX | XXX.XXX | XXX.XX | XX.X | XXX.X |
| Arm A | | | | | | | | | | | | | |
| Baseline | XXX | XXX.XX | XXX.XXX | XXX.XX | XX.X | XXX.X | XXX.XX | | | | | | |
| Cycle 1 Day 8 | XXX | XXX.XX | XXX.XXX | XXX.XX | XX.X | XXX.X | XXX.XX | XXX | XXX.XX | XXX.XXX | XXX.XX | XX.X | XXX.X |
| Cycle 1 Day 15 | XXX | XXX.XX | XXX.XXX | XXX.XX | XX.X | XXX.X | XXX.XX | XXX | XXX.XX | XXX.XXX | XXX.XX | XX.X | XXX.X |
| | XXX | XXX.XX | XXX.XXX | XXX.XX | XX.X | XXX.X | XXX.XX | XXX | XXX.XX | XXX.XXX | XXX.XX | XX.X | XXX.X |

- 1. Display the scheduled visits for this study.
- 2. Update the biomarker name in the title as appropriate.
- 3. Update the biomarker name in the first row of the table and unit as appropriate.

#### 5. NARRATIVE CRITERION

- Deaths within 30 days of last dose of study treatment
- Discontinuations of study treatment due to treatment-emergent AEs
- Treatment-emergent serious AEs
- Adverse events of clinical interest
  - Infusion-related reaction, Grade 3 or higher
  - Treatment-emergent Immune-related AE, Grade 3 or higher
  - Treatment-emergent infections/infestations, SAE or Grade 3 or higher
  - Treatment-emergent hemorrhage events, SAE or Grade 3 or higher
  - Treatment-emergent tumor lysis syndrome, SAE or Grade 3 or higher
  - New Malignancies
  - Treatment-emergent anaphylaxis or suspected anaphylaxis
- Treatment-emergent for subject who require the DIRA test result to confirm CR/sCR or treatment-emergent for subject who has earlier date of CR/sCR due to DIRA
- Treatment-emergent intravascular hemolysis
- Treatment-emergent interference with cross-matching and red blood cell antibody screening

# 6. PROGRAMMING CODE FOR STATISTICAL PROCEDURES (IF REQUIRED)

# 7. LIST OF POST HOC OUTPUT (IF REQUIRED)

| IDENTIFIER | OUTPUT TITLE | ANALYSIS SET | TO DO | REFERENCE<br>LAYOUT |
|------------|--------------|--------------|-------|---------------------|

### 8. ADDITIONAL ANALYSIS/DEVIATION RULES

Please see DPS part 2.

## **REFERENCES**

- 1. Durie BG, Harousseau JL, Miguel JS, et al. International uniform response criteria for multiple myeloma. Leukemia. 2006;20(9):1467-1473.
- 2. Kumar S, Paiva B, Anderson KC et al. International Myeloma Working Group consensus criteria for response and minimal residual disease assessment in multiple myeloma. Lancet Oncol. 2016;17(8):e328-46
- 3. Rajkumar SV, Harousseau JL, Durie B, et al. Consensus recommendations for the uniform reporting of clinical trials: report of the International Myeloma Workshop Consensus Panel 1. Blood. 2011;117(18):4691-4695

50